CLINICAL TRIAL: NCT03340181
Title: Study on the Myocardial Protective Effect of RIPC in Patients Undergoing OPCABG
Brief Title: Study on the Myocardial Protective Effect of Upper Limb Ischemic Preconditioning in Patients Undergoing Off-pump Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2017-100R
Record Dates: First submitted 2017-10-31; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: OPCABG
Keywords: RIPC, myocardial protective effect

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): 4 cycles of 5-min ischemia(using a blood pressure cuff inflated to 40mmHg over the patient's basic blood pressure) and 5-min repercussion are done on an upper limb.
  Interventions: Other: RIPC
- control (Sham Comparator): patient in control group using a blood pressure cuff on an upper limb without inflating
  Interventions: Other: RIPC

INTERVENTIONS:
Other: RIPC — 4 cycles of 5-min ischemia(using a blood pressure cuff inflated to 40mmHg over the patient's basic blood pressure) and 5-min repercussion are done on an upper limb before skin incision.

SUMMARY:
The purpose of the study was to verify the myocardial protective effect of RIPC in patients undergoing OPCABG.

DETAILED DESCRIPTION:
66 patients scheduled for OPCABG are randomly assigned to a RIPC group(n=33) or a control group(n=33). In the RIPC group, 4 cycles of 5-min ischemia(using a blood pressure cuff inflated to 40mmHg over the patient's basic blood pressure) and 5-min repercussion are done on an upper limb before skin incision. Patients in the control group wear the same cuff on an upper limb but no pressure is applied. Anesthetic and surgical techniques are standardized during the trial. Serum inflammatory cytokines and cardiac injury markers will be measured before and after surgery. Internal mammary artery and saphenous vein tissues will be collected during the surgery to assess hypoxia-inducible factor (Hif)-1a and other signalling proteins.

ELIGIBILITY:
Inclusion Criteria:

* serious changes in several coronary arteries that need to receive OPCABG
* NHYA II-III
* ASA II-III

Exclusion Criteria:

* LVEF< 35%
* acute myocardial infarction
* multiple organ dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
ICU staying time | average of 1 year
  the time patients spend in ICU after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hui-lin Wang, Phd, Principal Investigator — Fudan University
Locations (1):
- Huilin Wang, Shanghai, Shanghai Municipality, China